CLINICAL TRIAL: NCT04282187
Title: A Phase 2 Trial Investigating Decitabine in Combination With a JAK-Inhibitor as a Bridge to Allogeneic Hematopoietic Stem Cell Transplant in Patients With Accelerated/Blast Phase Myeloproliferative Neoplasms
Brief Title: Decitabine With Ruxolitinib, Fedratinib or Pacritinib for the Treatment of Accelerated/Blast Phase Myeloproliferative Neoplasms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1006644; NCI-2020-00749 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10419 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-02-19; First posted 2020-02-24 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Essential Thrombocythemia; Myelodysplastic Syndrome; Myelodysplastic/Myeloproliferative Neoplasm; Myeloproliferative Neoplasm; Myeloproliferative Neoplasm, Not Otherwise Specified; Polycythemia Vera; Primary Myelofibrosis; Secondary Myelofibrosis
Keywords: Myeloid and Monocytic Leukemia; Other Hematopoietic
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Thrombocythemia, Essential; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Myeloproliferative Disorders; Polycythemia Vera; Primary Myelofibrosis; Leukemia, Monocytic, Acute | interventions — Decitabine; Injections; ruxolitinib; fedratinib; 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (decitabine, ruxolitinib, fedratinib, pacritinib) (Experimental): Patients receive decitabine IV QD over 1 hour on days 1-10, and either ruxolitinib PO BID, fedratinib PO daily, or pacritinib PO BID on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood and bone marrow samples throughout the trial.
  Interventions: Drug: Decitabine; Drug: Ruxolitinib; Drug: Fedratinib; Other: Questionnaire Administration; Drug: Pacritinib; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 127716; 2''-Deoxy-5-azacytidine; 5-Aza-2''-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Drug: Ruxolitinib — Given PO
  Other Names: 941678-49-5; INCB-18424; Jakafi; Oral JAK Inhibitor INCB18424
Drug: Fedratinib — Given PO
  Other Names: 936091-26-8; SAR302503; TG101348
Other: Questionnaire Administration — Ancillary studies
Drug: Pacritinib — Given PO
  Other Names: 937272-79-2; Oral JAK2 Inhibitor SB1518; SB 1518; SB-1518; SB1518
Procedure: Biospecimen Collection — Undergo collection of blood and bone marrow samples
  Other Names: Biological Sample Collection

SUMMARY:
This phase II trial studies how well decitabine with ruxolitinib, fedratinib, or pacritinib works before hematopoietic stem cell transplant in treating patients with accelerated/blast phase myeloproliferative neoplasms (tumors). Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Ruxolitinib, fedratinib, and pacritinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving chemotherapy before a donor hematopoietic stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. The donated stem cells may also replace the patient's immune cells and help destroy any remaining cancer cells. Decitabine, with ruxolitinib, fedratinib, or pacritinib may work better than multi-agent chemotherapy or no pre-transplant therapy, in treating patients with accelerated/blast phase myeloproliferative neoplasms.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive decitabine intravenously (IV) once daily (QD) over 1 hour on days 1-10, and either ruxolitinib orally (PO) twice daily (BID), fedratinib PO daily, or pacritinib PO BID on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood and bone marrow samples throughout the trial.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* History of MPN as defined by the 2016 World Health Organization criteria, with now pathologically confirmed >= 5% blasts in the bone marrow or peripheral blood. Prior MPNs could include polycythemia vera, essential thrombocythemia, primary myelofibrosis, secondary myelofibrosis, MPN unclassifiable, MDS/MPN overlap
* Outside diagnostic material is acceptable as long as peripheral blood and/or bone marrow slides are reviewed at the study institution by pathology. Flow cytometric analysis of peripheral blood and/or bone marrow should be performed according to institutional practice guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 or Karnofsky >= 60%
* Serum creatinine clearance >= 50 ml/min calculated by the Cockcroft-Gault Equation (assessed within 14 days of study day 1)
* Total bilirubin =< 3 unless due to Gilbert's disease or hemolysis (total bilirubin > 3 is allowable if thought due to Gilbert's disease, hemolysis, or MPN disease) (assessed within 14 days of study day 1)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 3 x upper limit of normal (ULN) unless thought to be due to MPN disease process (AST/ALT > 3 is allowable if thought due to MPN disease) (assessed within 14 days of study day 1)
* For patient receiving fedratinib, thiamine level should be above the laboratory lower limit of normal (>= 70 nmol/L in the University of Washington [UW]/Seattle Cancer Care Alliance [SCCA] lab). If it is low, it may be repleted but should be rechecked and demonstrated to normalize prior to initiation of therapy
* Patient is considered a potential transplant candidate. The attending/treating physician will determine transplant candidacy at the time of consent
* The use of hydroxyurea prior to study registration is allowed. Patients with symptoms/signs of hyperleukocytosis, white blood count (WBC) > 100,000/uL, or with concern for other complications of high tumor burden or leukostasis (e.g. hypoxia, disseminated intravascular coagulation) can be treated with leukapheresis or may receive up to 2 doses of cytarabine (up to 500 mg/m^2 /dose) anytime prior to enrollment
* Capable of providing valid informed consent

Exclusion Criteria:

* Previous treatment with chemotherapy (e.g. hypomethylating agents or cytarabine-based regimens) for MPN with >= 5% blasts in the blood or marrow. Prior temporary measures to control blood counts is allowed. Prior treatment with hydroxyurea, interferons or JAK inhibitor therapy is allowed
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with anti-microbials and/or controlled or stable (e.g. if specific, effective therapy is not available/feasible or desired [e.g. chronic viral hepatitis, human immunodeficiency virus (HIV)])
* Known hypersensitivity to any study drug
* Females who are pregnant or breastfeeding
* Treatment with any other anti-MDS/leukemia investigational agent within 2 weeks of start of study drugs
* For patients planning to receive fedratinib: concurrent use of strong and moderate CYP3A4 inducers or dual CYP3A4 and CYP2C19 inhibitors that cannot be discontinued
* For patients planned to receive ruxolitinib AND platelets < 50,000/mm^2: concurrent use of a strong CYP3A4 inhibitor that cannot be discontinued
* For patients planned to receive pacritinib, corrected QT interval (QTc) > 480 msec (changing of medications/supplementing electrolytes is allowed to determine if this helps QTc reduce to < 480 msec)
* For patients planned to receive pacritinib, concurrent use of medications that are CYP1A2, CYP3A4, P-gp, BCRP, OCT1 substrates that cannot be discontinued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2026-11-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients enrolled who receive hematopoietic stem cell transplantation (HCT) | Up to 5 years

SECONDARY OUTCOMES:
Time from diagnosis of myeloproliferative neoplasm (MPN)-accelerated phase (AP)/blast phase (BP) to day 0 of HCT | Up to day 0 of HCT
  Estimated as a simple proportion and informally compared to rates seen historically among patients treated with multi-agent chemotherapy or no pre-HCT therapy.
Remission rate | At day 100
  Assessed via the Mascarenhas criteria. Estimated as a simple proportion and informally compared to rates seen historically among patients treated with multi-agent chemotherapy or no pre-HCT therapy.
Overall survival | From day 0 of HCT, assessed until 12 months post HCT
  Estimated as a simple proportion and informally compared to rates seen historically among patients treated with multi-agent chemotherapy or no pre-HCT therapy.
Relapse-free survival | From day 0 of HCT, assessed until 12 months post HCT
  Estimated as a simple proportion and informally compared to rates seen historically among patients treated with multi-agent chemotherapy or no pre-HCT therapy.
Mutational profiling | Up to 5 years
  Mutational data will be descriptive. The study team will record mutations found on the next generation of sequencing assays and will watch how these profiles change over time
Response rates regardless of transplant status | From day 1 of study treatment, assessed up to 5 years
  Assessed via Mascarenhas criteria. Estimated as a simple proportion and informally compared to rates seen historically among patients treated with multi-agent chemotherapy or no pre-HCT therapy.
Overall survival regardless of transplant status | From day 1 of study treatment, assessed up to 5 years
  Estimated as a simple proportion and informally compared to rates seen historically among patients treated with multi-agent chemotherapy or no pre-HCT therapy.
Relapse-free survival regardless of transplant status | From day 1 of study treatment, assessed up to 5 years
  Estimated as a simple proportion and informally compared to rates seen historically among patients treated with multi-agent chemotherapy or no pre-HCT therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Halpern, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No